CLINICAL TRIAL: NCT06405802
Title: Face-to-Face and Technology-Used Balance, Mobility and Strength Assessment in Patients With Low Back Pain
Brief Title: Comparison of Technology-assisted and Face-to-face Assessment in Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Bozyaka Training and Research Hospital (Other); Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Muhammed Zahid Uz, Lecturer, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022/142
Record Dates: First submitted 2024-05-04; First posted 2024-05-08 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Low Back Pain
Keywords: tele-evaluation; Low Back Pain; Face to face evaluation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-evulation (Experimental): Face-to-face tests will be recorded by video and re-evaluation will be made over the video by another person who has not performed the tests. During technology-based remote evaluations, the evaluator will monitor the tests simultaneously via video. During technology-based remote evaluations, video recording will be made and a re-evaluation will be made over the video by another person who has not performed the tests.
  Interventions: Other: Tele-evaluation
- Face-to face evulation (Experimental): Face-to-face applications were carried out with individuals with low back pain who came to Bozyaka Training and Research Hospital and volunteered to participate in the study.
  Interventions: Other: Tele-evaluation

INTERVENTIONS:
Other: Tele-evaluation — Evaluations will be carried out in two different environments: face-to-face in the clinic and remotely using technology. Face-to-face applications and remote evaluations using technology will be repeated once. Face-to-face applications will be made to individuals with low back pain who come to Bozyaka Training and Research Hospital and volunteer to participate in the study. Then, patients will be video-called at home, asked to perform the tests twice as taught, and recorded as a video.
  Other Names: Face to face evaluation

SUMMARY:
Although the concepts of telemedicine and tele-rehabilitation have been frequently emphasized in recent years, the evaluation part remains inadequate. There is no study investigating remote technology-based balance, mobility and strength assessments in patients with low back pain. Therefore, the aim of the study is; It is the examination of face-to-face and technology-based remote balance, mobility and strength assessment in patients with low back pain.

ELIGIBILITY:
Inclusion criteria

* Those over the age of 18
* People who can read and write
* Patients who have not undergone surgery
* Those whose body mass index is less than 30 m2/kg
* Volunteering to participate in the study

Exclusion criteria

* Patients who underwent surgery due to disc herniation
* Having any spinal pathology
* Having an uncontrolled neurological and metabolic disease
* Having a spinal deformity such as scoliosis or kyphosis
* Those with serious orthopedic, vascular, neurological or psychiatric problems that affect balance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Oswestry disability index | An evaluation was made once at the beginning of the research.
  The Oswestry Disability Questionnaire is a self-assessment tool that allows patients to assess the various constraints encountered during their daily activities. Utilizing a comprehensive scoring system ranging from 0 to 100, higher scores on the questionnaire indicate a heightened level of disability.
Timed-up and go test | An evaluation was made once at the beginning of the research.
  Simmonds et al. (1998) researched to ascertain the reliability of this test in swiftly and practically demonstrating functional status among patients with low back pain. The assessment involves the patient transitioning from seated to standing, traversing a 3-meter-long path, executing a turn, and returning to a seated posture. The duration of this performance is meticulously recorded
Single Leg Stance Test | An evaluation was made once at the beginning of the research.
  This examination, focused on assessing balance and static standing capacity, also offers insights into individuals' susceptibility to falls. During the evaluation process, participants were instructed to elevate their foot on their unaffected side and sustain this position for as long as possible. The termination of the test was determined by either contact of the free leg with the ground or a notable increase in arm oscillations
Thirty Second Chair Stand Test | An evaluation was made once at the beginning of the research.
  The Thirty Second Chair Stand Test is a validated and reliable assessment modality to gauge lower extremity strength (7). During the administration of this test, participants were tasked with repeatedly rising from and sitting back down on a chair within a 30-second timeframe, with the total number of repetitions recorded. A chair with a standardized sitting height of 43 cm was utilized for the assessments, and for safety precautions, it was positioned against a wall.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Zahid Uz, Master, Study Chair — Izmir Katip Çelebi University
Locations (1):
- Izmir Kâtip Çelebi University Vocational School of Health Services, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We aim to turn our research into an article and publish it in scientific journals.